CLINICAL TRIAL: NCT04031781
Title: The Role of Left Prefrontal Transcranial Magnetic Stimulation in Episodic Migraine Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Emara, Assistant professor of neurology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU 1171/2012
Record Dates: First submitted 2019-07-20; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Episodic Migraine; Prophylaxis
Keywords: rTMS = repetitive transcranial magnetic stimulation; LDLPFC = Left dorsolateral prefrontal cortex; HIT 6 = Headache Impact test; NPRS = Numeric Pain Rating Scale; ICHD = The international classfication of Headache disorder; MT= Motor threshold
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving repetitive transcranial magnetic stimulation (rTMS) (Active Comparator): This group received 5 rTMS sessions, delivered over one week over the left dorsolateral prefrontal cortex (LDLPFC ) at 5-Hz frequency and 100% motor threshold intensity.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS) 100% motor threshold
- Group receiving placebo rTMS (Placebo Comparator): This group received Placebo rTMS was given with the same stimulation frequency at a fixed intensity of 50% of the machine output
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS) 50% motor threshold

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) 100% motor threshold — Each rTMS session consisted of a single train of 900 total pulses over 3 minutes duration.
  Arms: Receiving repetitive transcranial magnetic stimulation (rTMS)
Device: repetitive transcranial magnetic stimulation (rTMS) 50% motor threshold — Each rTMS session consisted of a single train of 900 total pulses over 3 minutes duration.
  Arms: Group receiving placebo rTMS

SUMMARY:
The aim of the study was to examine the prophylactic role of repetitive transcranial magnetic stimulation (rTMS) on the frequency, and severity of migraine attacks in episodic migraineurs who failed medical treatment.

A group received 5 rTMS sessions, delivered over one week. Each rTMS session consisted of a single train of 900 total pulses over 3 minutes duration given at 5-Hz frequency and 100% motor threshold intensity and the placebo group received rTMS with the same stimulation frequency at a fixed intensity of 50% of the machine output

ELIGIBILITY:
Inclusion Criteria:

* cases diagnosed as episodic migraine with or without aura according to the ICHD 3rd edition
* With a headache frequency of 4-14 per month for the last six months
* Patients who had either an unsatisfactory response, declined or were intolerant to at least two prophylactic medications.

Exclusion Criteria:

* Patients with past family history of seizures
* Other chronic pain disorders
* Severe depression (Beck Depression Inventory of 30 or more)
* Other significant neurologic or psychiatric diagnosis including substance misuse
* Metal implants in the head
* Pregnant or breastfeeding ladies
* Prior experience with TMS

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-08-20 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Migraine attack frequency | 2 months
  The primary outcome measure was defined as the reduction of number of migraine attacks by at least 50% after rTMS sessions.

SECONDARY OUTCOMES:
Migraine days | 2 months
  Number of days that the migraine attack lasts in
Migraine attack severity | 2 months
  The intensity of pain that was assessed using the zero to ten Numeric Pain Rating Scale (NPRS)
Functional disability | 2 months
  Functional disability was measured using the HIT-6 score. Severe HIT-6 was defined as a score of 60 or more. A clinically significant change in the HIT-6 was defined as a change of five points or more.
Use of abortive pills | 2 months
  Number of pills used per month